CLINICAL TRIAL: NCT02640300
Title: Switching Antipsychotics: Abrupt Discontinuation Versus Overlap
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: The Ian Douglas Bebensee Foundation (Unknown)
Responsible Party: Principal Investigator, Gary Remington, Professor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4962
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: antipsychotics, clozapine, schizophrenia, switching strategy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate discontinuation group (Experimental): The antipsychotic drugs that patients took at baseline were prepared in unmarked capsules, with the dose adjusted to provide a 25% reduction weekly over the next 3 weeks. The dose tapering schedule was as follows: 3 capsules at baseline, 2 capsules at week 1, 1 capsule at week 2, and 0 capsules at week 3. All capsules contained placebo (i.e., the antipsychotic drugs were abruptly discontinued). Clozapine was gradually increased to 300 mg/day according to the following schedule: 12.5 mg/day at day 0 and increased by 25 mg/day to 300 mg/day at day 12, with this dose maintained for three weeks and thereafter adjusted according to clinical judgment. Concomitant medications were kept constant throughout the study period.
  Interventions: Drug: Clozapine
- Gradual discontinuation group (Experimental): The antipsychotic drugs that patients took at baseline were prepared in unmarked capsules, with the dose adjusted to provide a 25% reduction weekly over the next 3 weeks. The dose tapering schedule was as follows: 3 capsules at baseline, 2 capsules at week 1, 1 capsule at week 2, and 0 capsules (i.e., the antipsychotic drugs were discontinued) at week 3. Clozapine was gradually increased to 300 mg/day according to the following schedule: 12.5 mg/day at day 0 and increased by 25 mg/day to 300 mg/day at day 12, with this dose maintained for three weeks and thereafter adjusted according to clinical judgment. Concomitant medications were kept constant throughout the study period.
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine — Switching to clozapine with immediate or gradual antipsychotic discontinuation
  Other Names: Clozaril

SUMMARY:
Clozapine has been demonstrated to be clinically superior to other antipsychotics in treatment-resistant schizophrenia (TRS), and is positioned as such in treatment guidelines. Because it is relegated to use in TRS, guidelines require that it only be used after other antipsychotics have failed; accordingly, clinicians routinely contend with stopping the previous antipsychotic in making the switch to clozapine. Perhaps because of its numerous and potentially severe side effects, the issue of clozapine titration has frequently been addressed, although to our knowledge no study has, as of yet, assessed the comparability of gradual vs. immediate antipsychotic discontinuation in switching to clozapine. To address the gap in knowledge specific to clozapine, the investigators conducted a pilot, 8-week, double-blind, randomized controlled trial examining immediate vs. gradual antipsychotic discontinuation in patients with schizophrenia undergoing a switch to clozapine.

DETAILED DESCRIPTION:
Clozapine has been demonstrated to be clinically superior to other antipsychotics in treatment-resistant schizophrenia (TRS), and is positioned as such in treatment guidelines. Because it is relegated to use in TRS, guidelines require that it only be used after other antipsychotics have failed; accordingly, clinicians routinely contend with stopping the previous antipsychotic in making the switch to clozapine. Perhaps because of its numerous and potentially severe side effects, the issue of clozapine titration has frequently been addressed, although to our knowledge no study has, as of yet, assessed the comparability of gradual vs. immediate antipsychotic discontinuation in switching to clozapine.

While the question has not been asked vis-à-vis clozapine, there have been several studies examining gradual vs. immediate antipsychotic discontinuation in switching antipsychotics. Immediate antipsychotic discontinuation is associated with the following risks: (1) withdrawal/discontinuation symptoms or rebound syndromes related to cholinergic, histaminergic, and serotonergic activity; (2) supersensitivity syndromes (e.g., withdrawal dyskinesia, supersensitivity psychosis); and (3) exacerbation/re-emergence of symptoms secondary to diminished response with newly introduced antipsychotic. On the other hand, gradual antipsychotic discontinuation is associated with the risk of worsening/emergent side effects. This said, all of the studies, including one meta-analysis, report no differences in efficacy and safety between immediate and gradual discontinuation strategies in antipsychotic switching. However, it should be also noted that all of the studies were conducted under an open-label design or a single-blind design.

To address the gap in knowledge specific to clozapine, the investigators conducted a pilot, 8-week, double-blind, randomized controlled trial examining immediate vs. gradual antipsychotic discontinuation in patients with schizophrenia undergoing a switch to clozapine.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of schizophrenia or schizoaffective disorder based on the Structured Clinical Interview for DSM-IV (SCID-I)
* Candidacy for a trial of clozapine, defined as an inadequate clinical response to ≥ two antipsychotics (detailed in a pivotal clozapine study) and/or intolerable side effects

Exclusion Criteria:

* Active substance use disorder; inability to undergo a trial of clozapine for medical reasons (e.g., myeloproliferative disorder or history of drug-induced granulocytopenia)
* Evidence of significant nonadherence, defined as ≤75% adherence following patient interview, review of records, and discussion with treating physician and caregivers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 1999-05; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change in the Brief Psychiatric Rating Scale (BPRS) total scores from baseline to 8 weeks | 0 and 8 weeks

SECONDARY OUTCOMES:
Change in the Simpson-Angus Scale (SAS) total scores from baseline to 8 weeks | 0 and 8 weeks
Change in the Barnes Akathisia Rating Scale (BARS) total scores from baseline to 8 weeks | 0 and 8 weeks
Change in the Abnormal Involuntary Movement Scale (AIMS) overall severity scores from baseline to 8 weeks | 0 and 8 weeks
Change in the UKU Side Effect Rating Scale (UKU) subscale average scores from baseline to 8 weeks | 0 and 8 weeks
Change in the Clinical Global Impression - Severity scale (CGI-S) scores from baseline to 8 weeks | 0 and 8 weeks
Change in the Calgary Depression Scale for Schizophrenia (CDSS) total scores from baseline to 8 weeks | 0 and 8 weeks
Change in the Drug Attitude Inventory (DAI-10) total scores from baseline to 8 weeks | 0 and 8 weeks
Change in the Schedule for the Assessment of Insight (SAI) total scores from baseline to 8 weeks | 0 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Remington, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azorin JM, Spiegel R, Remington G, Vanelle JM, Pere JJ, Giguere M, Bourdeix I. A double-blind comparative study of clozapine and risperidone in the management of severe chronic schizophrenia. Am J Psychiatry. 2001 Aug;158(8):1305-13. doi: 10.1176/appi.ajp.158.8.1305. PMID 11481167
- [Background] Chakos M, Lieberman J, Hoffman E, Bradford D, Sheitman B. Effectiveness of second-generation antipsychotics in patients with treatment-resistant schizophrenia: a review and meta-analysis of randomized trials. Am J Psychiatry. 2001 Apr;158(4):518-26. doi: 10.1176/appi.ajp.158.4.518. PMID 11282684
- [Background] Lewis SW, Barnes TR, Davies L, Murray RM, Dunn G, Hayhurst KP, Markwick A, Lloyd H, Jones PB. Randomized controlled trial of effect of prescription of clozapine versus other second-generation antipsychotic drugs in resistant schizophrenia. Schizophr Bull. 2006 Oct;32(4):715-23. doi: 10.1093/schbul/sbj067. Epub 2006 Mar 15. PMID 16540702
- [Background] McEvoy JP, Lieberman JA, Stroup TS, Davis SM, Meltzer HY, Rosenheck RA, Swartz MS, Perkins DO, Keefe RS, Davis CE, Severe J, Hsiao JK; CATIE Investigators. Effectiveness of clozapine versus olanzapine, quetiapine, and risperidone in patients with chronic schizophrenia who did not respond to prior atypical antipsychotic treatment. Am J Psychiatry. 2006 Apr;163(4):600-10. doi: 10.1176/ajp.2006.163.4.600. PMID 16585434
- [Background] Souza JS, Kayo M, Tassell I, Martins CB, Elkis H. Efficacy of olanzapine in comparison with clozapine for treatment-resistant schizophrenia: evidence from a systematic review and meta-analyses. CNS Spectr. 2013 Apr;18(2):82-9. doi: 10.1017/S1092852912000806. Epub 2012 Dec 20. PMID 23253621
- [Background] Warnez S, Alessi-Severini S. Clozapine: a review of clinical practice guidelines and prescribing trends. BMC Psychiatry. 2014 Apr 7;14:102. doi: 10.1186/1471-244X-14-102. PMID 24708834
- [Background] Collins EJ, Lalonde P, Jones BD, Addington D, MacCrimmon DJ, MacEwan GW, Teehan MD. Clozapine in the treatment of refractory schizophrenia: Canadian policies and clinical guidelines. Can J Psychiatry. 1992 Sep;37(7):482-96. doi: 10.1177/070674379203700704. English, French. PMID 1423146
- [Background] Devinsky O, Honigfeld G, Patin J. Clozapine-related seizures. Neurology. 1991 Mar;41(3):369-71. doi: 10.1212/wnl.41.3.369. PMID 2006003
- [Background] Ifteni P, Nielsen J, Burtea V, Correll CU, Kane JM, Manu P. Effectiveness and safety of rapid clozapine titration in schizophrenia. Acta Psychiatr Scand. 2014 Jul;130(1):25-9. doi: 10.1111/acps.12241. Epub 2013 Dec 20. PMID 24354448
- [Background] Pacia SV, Devinsky O. Clozapine-related seizures: experience with 5,629 patients. Neurology. 1994 Dec;44(12):2247-9. doi: 10.1212/wnl.44.12.2247. PMID 7991106
- [Background] Ronaldson KJ, Fitzgerald PB, Taylor AJ, Topliss DJ, Wolfe R, McNeil JJ. Rapid clozapine dose titration and concomitant sodium valproate increase the risk of myocarditis with clozapine: a case-control study. Schizophr Res. 2012 Nov;141(2-3):173-8. doi: 10.1016/j.schres.2012.08.018. Epub 2012 Sep 23. PMID 23010488
- [Background] Kinon BJ, Basson BR, Gilmore JA, Malcolm S, Stauffer VL. Strategies for switching from conventional antipsychotic drugs or risperidone to olanzapine. J Clin Psychiatry. 2000 Nov;61(11):833-40. doi: 10.4088/jcp.v61n1105. PMID 11105736
- [Background] Lee CT, Conde BJ, Mazlan M, Visanuyothin T, Wang A, Wong MM, Walker DJ, Roychowdhury SM, Wang H, Tran PV. Switching to olanzapine from previous antipsychotics: a regional collaborative multicenter trial assessing 2 switching techniques in Asia Pacific. J Clin Psychiatry. 2002 Jul;63(7):569-76. doi: 10.4088/jcp.v63n0706. PMID 12143912
- [Background] Casey DE, Carson WH, Saha AR, Liebeskind A, Ali MW, Jody D, Ingenito GG; Aripiprazole Study Group. Switching patients to aripiprazole from other antipsychotic agents: a multicenter randomized study. Psychopharmacology (Berl). 2003 Apr;166(4):391-9. doi: 10.1007/s00213-002-1344-3. Epub 2003 Feb 28. PMID 12610718
- [Background] Weiden PJ, Simpson GM, Potkin SG, O'Sullivan RL. Effectiveness of switching to ziprasidone for stable but symptomatic outpatients with schizophrenia. J Clin Psychiatry. 2003 May;64(5):580-8. doi: 10.4088/jcp.v64n0514. PMID 12755663
- [Background] Ganguli R, Brar JS, Mahmoud R, Berry SA, Pandina GJ. Assessment of strategies for switching patients from olanzapine to risperidone: a randomized, open-label, rater-blinded study. BMC Med. 2008 Jun 30;6:17. doi: 10.1186/1741-7015-6-17. PMID 18590519
- [Background] Pae CU, Serretti A, Chiesa A, Mandelli L, Lee C, Lee C, Kim J, De Ronchi D, Paik IH. Immediate versus gradual suspension of previous treatments during switch to aripiprazole: results of a randomized, open label study. Eur Neuropsychopharmacol. 2009 Aug;19(8):562-70. doi: 10.1016/j.euroneuro.2009.04.002. Epub 2009 May 12. PMID 19442491
- [Background] Stip E, Zhornitsky S, Potvin S, Tourjman V. Switching from conventional antipsychotics to ziprasidone: a randomized, open-label comparison of regimen strategies. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Aug 16;34(6):997-1000. doi: 10.1016/j.pnpbp.2010.05.010. Epub 2010 May 12. PMID 20470848
- [Background] Weiden PJ, Citrome L, Alva G, Brams M, Glick ID, Jackson R, Mattingly G, Kianifard F, Meng X, Pestreich L, Hochfeld M, Winseck A. A trial evaluating gradual- or immediate-switch strategies from risperidone, olanzapine, or aripiprazole to iloperidone in patients with schizophrenia. Schizophr Res. 2014 Mar;153(1-3):160-8. doi: 10.1016/j.schres.2013.11.042. Epub 2014 Feb 12. PMID 24529610
- [Background] Cerovecki A, Musil R, Klimke A, Seemuller F, Haen E, Schennach R, Kuhn KU, Volz HP, Riedel M. Withdrawal symptoms and rebound syndromes associated with switching and discontinuing atypical antipsychotics: theoretical background and practical recommendations. CNS Drugs. 2013 Jul;27(7):545-72. doi: 10.1007/s40263-013-0079-5. PMID 23821039
- [Background] Remington G, Chue P, Stip E, Kopala L, Girard T, Christensen B. The crossover approach to switching antipsychotics: what is the evidence? Schizophr Res. 2005 Jul 15;76(2-3):267-72. doi: 10.1016/j.schres.2005.01.009. PMID 15949658
- [Background] Kane J, Honigfeld G, Singer J, Meltzer H. Clozapine for the treatment-resistant schizophrenic. A double-blind comparison with chlorpromazine. Arch Gen Psychiatry. 1988 Sep;45(9):789-96. doi: 10.1001/archpsyc.1988.01800330013001. PMID 3046553
- [Derived] Takeuchi H, Lee J, Fervaha G, Foussias G, Agid O, Remington G. Switching to Clozapine Using Immediate Versus Gradual Antipsychotic Discontinuation: A Pilot, Double-Blind, Randomized Controlled Trial. J Clin Psychiatry. 2017 Feb;78(2):223-228. doi: 10.4088/JCP.15m10286. PMID 28234436
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research